CLINICAL TRIAL: NCT02448615
Title: A Longitudinal Birth Cohort Study in Coast Province, Kenya
Brief Title: Birth Cohort in Coast Province, Kenya
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: March of Dimes (Other); Grand Challenges Canada (Other); Aga Khan University (Other)
Responsible Party: Principal Investigator, Shaun Morris, Clinician-Scientist, The Hospital for Sick Children
Other Study IDs: 1000047574
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Mortality; Morbidity; Child Development; Child Behaviour
Keywords: Kenya; Cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Birth Cohort: The cohort will comprise approximately 1500 pregnant women and their unborn babies, enrolled to participate in the control arm of a cluster-randomized controlled intervention trial (NCT02208960).

SUMMARY:
In 2010, 7.6 million children under the age of five died worldwide and yet the causes of only 2.7% (0.205 million) of these deaths were medically certified. A thorough understanding of the causes of child mortality is necessary to guide research efforts aimed at tackling this important global health problem. Prospective birth cohort studies present an opportunity to examine the relationships between early-life exposures and multiple health and non-health related outcomes including death, illness, and socioeconomic factors. In this study, the investigators will provide insight into the underlying causes of child mortality by collecting data on early-life exposures and health and non-health related outcomes in the first year of life.

DETAILED DESCRIPTION:
In 2010, 7.6 million children under the age of five died worldwide, mainly from preventable and treatable conditions (Liu et al., 2012). Notably, the burden of under-five mortality varies dramatically by country. The majority of child deaths are seen in Africa (3.6 million) and southeast Asia (2.1 million deaths), compared to 0.16 million and 0.28 million under-five deaths in Europe and the Americas, respectively (Liu et al., 2012). In Kenya, over 120,000 under-5 deaths were estimated in 2010 and approximately 35% of these deaths occurred in the neonatal period.

A thorough understanding of the etiology of child mortality is necessary to guide research efforts aimed at tackling this important global health problem. Importantly, in 2010, the causes of only 2.7% (0.205 million) of all deaths in children under the age of five were medically certified (Liu et al., 2012), highlighting the need to gather data on the causes of mortality.

Prospective longitudinal birth cohort studies present an opportunity to examine temporal relationships between early-life exposures (i.e. prenatal, pregnancy, and early postnatal exposures) and multiple health and non-health related outcomes including mortality, morbidity, and socioeconomic circumstances. It is well documented that exposures that occur early in life, including genetic, environmental, socioeconomic, and lifestyle factors, may have long-lasting effects on growth, development, and health outcomes throughout an individual's entire life course (Lynch & Smith, 2005). Thus, data on exposures during pregnancy and early childhood are valuable and may provide clues to the etiology of long-term outcomes.

Additional value can be gained through cross-cohort collaborations and comparisons (Larsen et al., 2013)(Paternoster et al., 2012)(Brion et al., 2011). Notably, by pooling data from multiple cohort studies, causal inferences can be made with greater confidence. For example, if a similar relationship is observed across multiple populations, each with their own distinct set of confounding variables, it is less likely that the observed association is being driven by confounders. Similarly, cross-cohort comparisons enable researchers to investigate patterns associated with health, social, and economic outcomes in distinct regions of the world. These types of analyses may provide valuable insight into the underlying causes of global health inequalities.

The objective of this study is to implement a longitudinal prospective birth cohort study in Kenya to obtain extensive information on early-life exposures and health and non-health related outcomes in the first year of life.

ELIGIBILITY:
Inclusion Criteria:

i. All pregnant women and their home- or facility-born live newborns that consent to participate in the control arm of the study "An integrated toolkit to save newborn lives and brains in Kenya" (NCT02208960) will be eligible for this study. The maternal inclusion criteria will be:

1. All pregnant women in parts of study clusters covered by CHW program and their home- or facility-born live newborns.
2. Mothers intending to maintain residence in study area for first 12 months of newborn's life.

Exclusion Criteria:

i. Did not consent to participate in the control arm of "An integrated toolkit to save newborn lives and brains in Kenya" (NCT02208960).

ii. Failure to provide consent to enroll in this study.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pregnant women (and their unborn newborns) who consent to participate in the control arm of the previously approved trial "An integrated toolkit to save newborn lives and brains in Kenya" (NCT02208960) will be eligible for enrollment in this study. At the time of consent, participants will be informed that they are free to consent to the neonatal kit trial without consenting to the birth cohort study.
Sampling Method: Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Child mortality within the first year of life | 12 months (Day 3 of life, Month 6 of life, Month 12 of life)
  Death from any cause within the first year of life will be assessed by questionnaire.

SECONDARY OUTCOMES:
Morbidity within the first year of a child's life | 12 months (Day 3 of life, Month 6 of life, Month 12 of life)
  The most common types of illness within the first year of a child's life will be assessed by questionnaire.
Development/behaviour of children aged 6 and 12 months in the Coast Province, Kenya | Month 6 of life, Month 12 of life
  Assessed by questionnaire (month 6) and questionnaire and Kilifi Developmental Inventory at month 12. Linear growth and weight are collected at day 3, month 6 and month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Shaun K Morris, MD, MPH, Principal Investigator — The Hospital for Sick Children; Robert Armstrong, MD, PhD, Principal Investigator — Aga Khan University
Locations (2):
- Kenya (2):
  - Community, Kwale, Coast Province
  - Aga Khan University, Nairobi

REFERENCES:
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] Lynch J, Smith GD. A life course approach to chronic disease epidemiology. Annu Rev Public Health. 2005;26:1-35. doi: 10.1146/annurev.publhealth.26.021304.144505. PMID 15760279
- [Background] Larsen PS, Kamper-Jorgensen M, Adamson A, Barros H, Bonde JP, Brescianini S, Brophy S, Casas M, Charles MA, Devereux G, Eggesbo M, Fantini MP, Frey U, Gehring U, Grazuleviciene R, Henriksen TB, Hertz-Picciotto I, Heude B, Hryhorczuk DO, Inskip H, Jaddoe VW, Lawlor DA, Ludvigsson J, Kelleher C, Kiess W, Koletzko B, Kuehni CE, Kull I, Kyhl HB, Magnus P, Momas I, Murray D, Pekkanen J, Polanska K, Porta D, Poulsen G, Richiardi L, Roeleveld N, Skovgaard AM, Sram RJ, Strandberg-Larsen K, Thijs C, Van Eijsden M, Wright J, Vrijheid M, Andersen AM. Pregnancy and birth cohort resources in europe: a large opportunity for aetiological child health research. Paediatr Perinat Epidemiol. 2013 Jul;27(4):393-414. doi: 10.1111/ppe.12060. PMID 23772942
- [Background] Brion MJ, Zeegers M, Jaddoe V, Verhulst F, Tiemeier H, Lawlor DA, Smith GD. Intrauterine effects of maternal prepregnancy overweight on child cognition and behavior in 2 cohorts. Pediatrics. 2011 Jan;127(1):e202-11. doi: 10.1542/peds.2010-0651. Epub 2010 Dec 27. PMID 21187310
- [Background] Paternoster L, Standl M, Chen CM, Ramasamy A, Bonnelykke K, Duijts L, Ferreira MA, Alves AC, Thyssen JP, Albrecht E, Baurecht H, Feenstra B, Sleiman PM, Hysi P, Warrington NM, Curjuric I, Myhre R, Curtin JA, Groen-Blokhuis MM, Kerkhof M, Saaf A, Franke A, Ellinghaus D, Folster-Holst R, Dermitzakis E, Montgomery SB, Prokisch H, Heim K, Hartikainen AL, Pouta A, Pekkanen J, Blakemore AI, Buxton JL, Kaakinen M, Duffy DL, Madden PA, Heath AC, Montgomery GW, Thompson PJ, Matheson MC, Le Souef P; Australian Asthma Genetics Consortium (AAGC); St Pourcain B, Smith GD, Henderson J, Kemp JP, Timpson NJ, Deloukas P, Ring SM, Wichmann HE, Muller-Nurasyid M, Novak N, Klopp N, Rodriguez E, McArdle W, Linneberg A, Menne T, Nohr EA, Hofman A, Uitterlinden AG, van Duijn CM, Rivadeneira F, de Jongste JC, van der Valk RJ, Wjst M, Jogi R, Geller F, Boyd HA, Murray JC, Kim C, Mentch F, March M, Mangino M, Spector TD, Bataille V, Pennell CE, Holt PG, Sly P, Tiesler CM, Thiering E, Illig T, Imboden M, Nystad W, Simpson A, Hottenga JJ, Postma D, Koppelman GH, Smit HA, Soderhall C, Chawes B, Kreiner-Moller E, Bisgaard H, Melen E, Boomsma DI, Custovic A, Jacobsson B, Probst-Hensch NM, Palmer LJ, Glass D, Hakonarson H, Melbye M, Jarvis DL, Jaddoe VW, Gieger C; Genetics of Overweight Young Adults (GOYA) Consortium; Strachan DP, Martin NG, Jarvelin MR, Heinrich J, Evans DM, Weidinger S; EArly Genetics & Lifecourse Epidemiology (EAGLE) Consortium. Meta-analysis of genome-wide association studies identifies three new risk loci for atopic dermatitis. Nat Genet. 2011 Dec 25;44(2):187-92. doi: 10.1038/ng.1017. PMID 22197932